CLINICAL TRIAL: NCT06295822
Title: The Effectiveness of Chinese Medicine Nuan-gong-ye on Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH112-REC2-063
Record Dates: First submitted 2024-02-25; First posted 2024-03-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Chinese Medicine; Primary Dysmenorrhea
Keywords: Chinese Medicine; Nuan-gong-ye; Primary dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nuan-gong-ye (Experimental)
  Interventions: Drug: Nuan-gong-ye
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nuan-gong-ye — In this study, the ingredients of nuan-gong-ye are myrrh, dragon's blood, yanhu tuber, white mustard seed, asarum root, argy wormwood leaf, holly oil, clove oil, cinnamon bark oil, glycerin, PEG400.
  Arms: Nuan-gong-ye
Other: Placebo — The placebo was 1/20 concentration of nuan-gong-ye plus glycerin and PEG400.
  Arms: Placebo

SUMMARY:
Primary dysmenorrhea is a common under-diagnosed complaint, with a prevalence of about 45-95% in women of childbearing age and about 10-25% in severe cases. Menstrual pain can be classified as primary or secondary. Primary menstrual pain is a crampy pain in the lower abdomen without any pelvic pathology, which usually occurs 6 to 12 months after the first menstruation. Primary menstrual pain is usually most severe on the first day of the menstrual cycle and lasts for 8 to 72 hours. The cause is still unknown, but studies suggest that it may be related to increased prostaglandins, which cause painful contractions of the uterus. The pain is often accompanied by other menstrual discomfort symptoms, including headache, breast tenderness, drowsiness, nausea, vomiting, constipation or diarrhea, and psychological anxiety, depression or irritability. In the case of secondary menstrual pain, there are clear pelvic pathologies, such as endometriosis, uterine fibroids, and pelvic inflammatory disease.

DETAILED DESCRIPTION:
In this study, the ingredients of nuan-gong-ye are myrrh, dragon's blood, yanhu tuber, white mustard seed, asarum root, argy wormwood leaf, holly oil, clove oil, cinnamon bark oil, glycerin, PEG400, while the placebo was 1/20 concentration of nuan-gong-ye plus glycerin and PEG400, all from the same batch. A bottle of nuan-gong-ye will be taken for HPLC fingerprint to examine its components. A total of 140 people will be divided randomly into two groups, of which the experimental group using nuan-gong-ye and the control group using a placebo. Four menstrual cycles of the clinical trial will be conducted after recruitment. The first menstrual cycle will be non-interventional, with subjects filling out Basic information sheet, Visual Analogue Scale (VAS), and Short Form McGill Pain Questionnaire (MPQ-SF). In the second to fourth menstrual cycles, two bottles of approximately 16 ml of nuan-gong-ye will be applied. During these three cycles, the application will begin five days before each menstrual period and end on the third day of the menstruation, with the VAS, McGill scale, and side effects questionnaire being completed. The skin should be dry before application. For each application of nuan-gong-ye or placebo, apply 10 circles clockwise from the navel to a circular area with a radius of 8 to 13 cm. The first application will be done after waking up, the second and third apply every five hours, and the fourth apply at bedtime, for a total of four applications a day. Other relief measures such as Chinese medicine, hot compresses, abdominal massage, acupuncture, and the use of other essential oils are prohibited during the research period, while painkillers are not.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 year-old women
* Regular menstrual cycle of 21-35 days, with menstruation lasting 3-7 days
* Dysmenorrhea started before the age of 20, and have menstrual pain every month
* No organic lesions on ultrasound within one year (either abdomen or vagina)
* VAS score above 4
* Agree to participate in the study and sign the consent form

Exclusion Criteria:

* Has used the same formula of Nuan-gong-ye before.
* Allergic to Nuan-gong-ye.
* Has abdominal wounds, infections, or skin diseases.
* Pregnant or planning to become pregnant within the next five months.
* Has taken traditional Chinese medicine or prescribed medication for menstrual pain by a Chinese medicine doctor in the past month.
* Has major illnesses defined by the Taiwan National Health Insurance Administration, such as cancer, heart disease, etc.
* Has mental illness or cognitive impairment and cannot independently fill out the questionnaire.
* Has a history of epilepsy or pelvic disorders.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 4 months
  The intensity of menstrual pain was measured by the Visual Analogue Scale (VAS). The VAS scale is a continuous horizontal line ten centimeters in length. The left end of the line, marked as 0, represents 'no pain,' while the right end, marked as 10, represents 'the most intense pain'. The VAS and McGill scales were used to assess the difference before and after each menstrual cycle.

SECONDARY OUTCOMES:
Short Form McGill Pain Questionnaire (MPQ-SF) | 4 months
  Pain perception was measured by the Short Form McGill Pain Questionnaire (MPQ-SF). The scale consists of 15 items, with scores ranging from 0 to 3 to assess the intensity of each pain. 0 represents 'none,' 1 represents 'mild pain,' 2 represents 'moderate pain,' and 3 represents 'severe pain.' The VAS and McGill scales were used to assess the difference before and after each menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No